CLINICAL TRIAL: NCT07349862
Title: THE IMPACT OF CANCER SCREENING TRAINING, CONDUCTED USING A CHATGPT-SUPPORTED FLIPPED LEARNING MODEL, ON NURSING STUDENTS' ACADEMIC KNOWLEDGE, LEARNING MOTIVATION, AND CLASSROOM ENGAGEMENT
Brief Title: Flipped Learning in Nursing Education
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Dilek Erden, Principal Investigator, Assistant Professor (Dr.), Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DERDEN-4
Record Dates: First submitted 2025-12-22; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Nursing Students; Education; Flipped Education Model
Keywords: learning motivation; classroom engagement; flipped learning; ChatGPT

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- ChatGPT Flipped Learning (Experimental): ChatGPT-Based Flıpped Learnıng Model
  Interventions: Other: ChatGPT-Based Flıpped Learning Model
- Control Group- Traditioanl Flipped Learning (Placebo Comparator): Traditional Flıpped Learnıng Model
  Interventions: Other: Traditional Flıpped Learning Model

INTERVENTIONS:
Other: ChatGPT-Based Flıpped Learning Model — Training group based on ChatGPT-based flipped learning model
  Arms: Intervention group- ChatGPT Flipped Learning
Other: Traditional Flıpped Learning Model — Training group based on traditional flipped learning model
  Arms: Control Group- Traditioanl Flipped Learning

SUMMARY:
This study aims to examine the effects of cancer screening training, conducted using a ChatGPT-based flipped learning model, on knowledge, learning motivation, and class participation.

DETAILED DESCRIPTION:
Methods: A randomized controlled trial was conducted with 46 intervention and 46 control groups. In the study, a training program based on traditional flipped learning and a ChatGPT-based flipped learning model for cancer screenings is applied. Data will be collected using the Knowledge Form, Cancer Screening Knowledge Scale, Higher Education Learning Motivation Scale, and Class Participation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Students who have taken courses in fundamentals of nursing, internal medicine nursing, physiology, pathology, and computer science, but have not taken a course in oncology nursing,
* Third-year students,
* Those who have voluntarily agreed to participate in the study.

Exclusion Criteria:

* Students who were not third-year students,
* Those who had not taken one of the following courses: fundamentals of nursing, internal medicine nursing, physiology, pathology, computer science, oncology nursing,
* Those who did not volunteer to participate in the research were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Cancer Screening Knowledge Scale | 4 weeks
  This scale consists of 25 items and 3 sub-dimensions. The sub-dimensions are not specifically named. The first sub-dimension contains 10 items (items 8, 17-23, 25, 28), the second sub-dimension contains 9 items (items 4, 5, 7, 10, 12, 13, 15, 16, 27), and the third sub-dimension contains 6 items (items 1-3, 9, 11, 24). The scale is a three-point rating scale. The scale is answered on a scale of 1 to 3, with "1: True, 2: False, 3: I don't know". When calculating the scale score, "True" answers are worth 1 point, and "False" and "I don't know" answers are worth 0 points. The lowest possible score on the scale is 0, and the highest is 25. When calculating the scale score, the three items with negative connotations (Items 2, 11, 24) should be reverse-coded. The order of the items on the scale is not important; researchers may use a mixed order. There is no cutoff point for the scale score.

SECONDARY OUTCOMES:
Learning Motivation Scale in Higher Education | 4 weeks
  The scale consisting of 23 items on a 3-point Likert scale, participants are given scores of Disagree (1), Don't Know (2), and Agree (3) for each question in the Learning Motivation Scale in Higher Education. The lowest possible score is 23 and the highest is 69. In the reliability studies of the scale, the Cronbach alpha coefficient of the learning objectives sub-dimension was calculated as 0.83, the avoidance objectives sub-dimension as 0.87, and the approach objectives sub-dimension as 0.82.

OTHER OUTCOMES:
Classroom Engagement Scale | 4 weeks
  The scale consisting of 15 items and 3 sub-dimensions on a 5-point Likert scale, participants are given scores for each question on a scale of 1 (Not Appropriate at all), 2 (Not Appropriate), 3 (Somewhat Appropriate), 4 (Appropriate), and 5 (Completely Appropriate). The scale includes sub-dimensions of Cognitive participation, Emotional participation, and Behavioral participation. In reliability studies of the scale, the Alpha value was found to be 0.93.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK ERDEN, Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I can share it with researchers who request it for reasonable reasons.